CLINICAL TRIAL: NCT05137990
Title: The Effects of High Intensity Exercise in Teens on Cognition
Brief Title: The HIIT Cognition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Britni Ryan Belcher, PhD, MPH, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS-21-00149
Record Dates: First submitted 2021-10-06; First posted 2021-11-30 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: High Intensity Interval Training; Overweight and Obesity; Metabolic Disease; Cognition
Keywords: High Intensity Interval Training; Physical Activity; Pediatric Obesity; Metabolic Disturbances; Mental Health
MeSH Terms: conditions — Overweight; Obesity; Metabolic Diseases; Motor Activity; Pediatric Obesity; Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to complete one of two conditions: 1) 14 weeks of a home-based virtual HIIT exercise intervention or 2) 14 weeks of a stretching intervention (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Exercise Intervention (Experimental): At home (N=12): Participants will complete an exercise session 3 times a week for 14 weeks. Each participant will receive a pre-assembled stationary bicycle to use to complete each session, an iPad to receive the intervention virtually from exercise trainers through Zoom, and a Fitbit to assess real-time heart rate.
  Interventions: Behavioral: HIIT Exercise Intervention
- Stretching Intervention (Placebo Comparator): At home (N=12): Participants will complete a stretching protocol 3 times a week for 14 weeks. Participants will be asked to complete weekly records of flexibility compliance.
  Interventions: Behavioral: Stretching Intervention

INTERVENTIONS:
Behavioral: HIIT Exercise Intervention — Exercise trainers will provide encouragement and supervision for exercise prescription adherence and youth will select an age-appropriate music playlist from Spotify to enhance enjoyment throughout each session. Each exercise session consists of a 5-minute warm-up (10% HRmax), followed by a 20-minute HIIT protocol. The 20-minute HIIT protocol consists of seven bouts of 1-min high intensity exercise (90% HRmax) followed by 2-min of active recovery (10% HRmax). Participants will be encouraged to complete each exercise session with at least 24 hours of rest between each session.
  Other Names: Exercise group
  Arms: HIIT Exercise Intervention
Behavioral: Stretching Intervention — This group will perform a home-based program of the same stretches utilized in the exercise group. The stretching protocol consists of one set of 4 static stretching exercises held for 30 seconds and performed 3 days/week. As flexibility exercises are low-intensity, low-impact and low-volume, minimal caloric expenditure is expected to be incurred. To increase compliance and aid in the standardization of the home-based stretching, participants will be provided a booklet of the flexibility exercises. Participants will be shown how to use the booklet and instructed in the stretching exercises by an exercise trainer prior to the intervention.
  Other Names: Control group
  Arms: Stretching Intervention

SUMMARY:
This pilot study is a randomized control trial to test the effects of a 14-week home-based virtual, interactive high intensity interval training (HIIT) exercise intervention on cardiometabolic and cognitive outcomes in sedentary youth with overweight/obesity during adolescence. All participants (N=24) will complete screening via phone to determine eligibility. Eligible participants will be randomized to receive a) 14 weeks of a home-based HIIT intervention delivered via iPad or b) 14 weeks of a stretching intervention (control group). Each participant will undergo an in-lab pre- and post-test visit, where they will complete a fasting blood draw, a fitness test, and various cognitive and mental health measures.

DETAILED DESCRIPTION:
Rationale: Existing literature supports the premise that physical activity (PA) has beneficial effects on cognitive function in youth, but prior studies have limitations, such as cross-sectional designs with limited insights on the intensity or duration of PA or the biological underpinnings linking physical activity and mental health and cognitive function in adolescents. A limited number of studies (and none in the U.S.) have evaluated the effects of HIIT on cognitive processes in youth, particularly in youth with overweight/obesity whose age-related declines in PA puts them at increased risk for poor outcomes. This study is particularly timely during the current COVID-19 related public health crisis because our HIIT exercise intervention is time efficient, delivered remotely, and completed using space-efficient equipment in the home.

Intervention: Participants (youth ages 12-16 years with overweight/obesity) will be randomly assigned to complete a) 14 weeks of a home-based virtual, interactive HIIT intervention or b) 14 weeks of a stretching intervention (control group).

Objectives/Purpose: The overall goal is to improve cognitive and cardiometabolic outcomes in youth with overweight/obesity by implementing an at-home HIIT intervention. The aims of this study are: 1) to determine the feasibility, acceptability, and efficacy of HIIT in adolescents with overweight/obesity, 2) to examine the effectiveness of HIIT on cognitive and mental health outcomes, and 3) to examine the effectiveness of HIIT on cardiometabolic health.

Study Population: This study will consist of youth ages 12-16 years with overweight/obesity (BMI >=85th percentile) who do not meet current PA guidelines.

Study Methodology: This pilot study is a randomized control trial to test the effects of a 14-week home-based virtual, interactive high intensity interval training (HIIT) exercise intervention on cardiometabolic and cognitive outcomes in sedentary youth with overweight/obesity during adolescence. All participants (N=24) will complete screening via phone to determine eligibility. Eligible participants will be randomized to receive a) 14 weeks of a home-based HIIT intervention delivered via iPad (HIIT group) or b) 14 weeks of a stretching intervention (control group).

Those randomized to the HIIT group will receive the intervention 3 times/week and will be given a pre-assembled stationary bicycle to use to complete each exercise session, an iPad to Zoom with the exercise trainers, and a Fitbit to assess real-time heart rate. Exercise trainers will provide encouragement and supervision for exercise prescription adherence and youth will select an age-appropriate music playlist from Spotify to enhance enjoyment throughout each session. Each exercise session consists of a 5-minute warm-up (10% HRmax), followed by a 20-minute HIIT protocol. The 20-minute HIIT protocol consists of seven bouts of 1-min high intensity exercise (90% HRmax) followed by 2-min of active recovery (10% HRmax). Participants will be encouraged to complete each exercise session with at least 24 hours of rest between each session.

Those randomized to the control group will perform a home-based program of the same stretches utilized in the exercise group. The stretching protocol consists of one set of 4 static stretching exercises held for 30 seconds and performed 3 days/week. As flexibility exercises are low-intensity, low-impact and low-volume, minimal caloric expenditure is expected to be incurred.

Study arms: Study participants will be randomly assigned to receive either the HIIT intervention (HIIT group) or receive the stretching intervention (control group).

Endpoints/Outcomes: The primary cognitive and mental health endpoints are: executive function, episodic memory, working memory, affect, mood, anxiety, stress, self-efficacy for PA, and PA enjoyment. The primary cardiometabolic endpoints are: glucose, insulin (to calculate Homeostatic Model Assessment for Insulin Resistance), IL-6, IL-1, TNF-a, and VEGF.

Statistical analyses: The populations for analyses include the full analytical dataset which consists of all randomized study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Typically developing youth.
2. Overweight/obese (BMI >= 85th percentile)
3. Does not meet current PA guidelines
4. Able and willing to complete HIIT exercise intervention.
5. Space for a stationary bike in the residence.

Exclusion Criteria:

1. Diagnoses of neurodevelopment or psychiatric disorders.
2. Diabetes, cardiovascular, pulmonary, or other significant medical problems.
3. Taking medications know to alter metabolism.
4. Allergy to metals.
5. Inability to participate in HIIT-based exercise or active involvement in sports/exercise programs.
6. Pregnancy.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Measures of intervention feasibility | 14 weeks
  percent of youth who complete an average of 70% of weekly minutes and percent of youth who attend 70% of exercise sessions
Measures of intervention efficacy | 14 weeks
  percent of sessions where youth achieve their target heart rate
Intervention Feasibility Measure | 14 weeks
  4-item scale with scores for each ranging from 1 to 5, higher scores indicate a better outcome for feasibility
Intervention Acceptability Measure | 14 weeks
  4-item scale with scores for each ranging from 1 to 5; higher scores indicate a better outcome for acceptability
Intervention Appropriateness Measure | 14 weeks
  4-item scale with scores for each ranging from 1 to 5; higher scores indicate a better outcome for appropriateness
Cognitive function measures | 14 weeks
  executive function, episodic and working memory tasks from NIH Toolbox, all age-adjusted T-scores
Positive and Negative Affect Scale for Children | 14 weeks
  10-item positive and negative affect scale with scores for each ranging from 0 to 5; higher scores indicate a worse outcome for negative affect and better outcome for positive affect
Profile of Mood States for Adolescents | 14 weeks
  24-item scale with each ranging from 0 to 4; higher scores indicate a worse mood outcome
State-Trait Anxiety Inventory for Children | 14 weeks
  20-item scale measuring acute and long-term anxiety, with a range from 20 to 80; higher scores indicate more anxiety
Perceived Stress Scale | 14 weeks
  10-item scale with each ranging from 0 to 4; higher scores indicate a worse stress outcome after reverse coding applicable items
Stress in Children Scale | 14 weeks
  21-item scale with each ranging from 0 to 4; higher scores indicate a worse stress outcome after reverse coding applicable items
Self-Efficacy for Physical Activity Scale | 14 weeks
  5-item scale with each ranging from 1 to 5; higher scores indicating a better self-efficacy for physical activity outcome
Physical Activity Enjoyment Scale | 14 weeks
  18-item scale with each ranging from 1 to 7; higher scores indicate a better physical activity enjoyment outcome after reverse coding applicable items
Glucose Sensitivity | 14 weeks
  glucose, insulin (to calculate Homeostatic Model Assessment for Insulin Resistance)
Markers of inflammation | 14 weeks
  interleukin-1 (IL-1), interleukin-6 (IL-6), tumor necrosis factor alpha (TNF-a), all in pg/mL
Vascular Endothelial-Derived Growth | 14 weeks
  vascular endothelial growth factor (VEGF) in pg/mL
Cardiorespiratory Fitness | 14 weeks
  maximal oxygen consumption (VO2max)
Blood Pressure | 14 weeks
  systolic and diastolic blood pressure
Body proportion | 14 weeks
  waist-to-height ratio
Body composition | 14 weeks
  percent body fat

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not intend to share IPD with other researchers outside of our study.